CLINICAL TRIAL: NCT05058755
Title: Efficacy and Safety of Tislelizumab Combined Treatment in Refractory Natural Killer/T-cell Lymphoma
Brief Title: Tislelizumab Combined Treatment in Refractory Extranodal NK/T-cell Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Rong Tao, MD, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHLSG-NK-1903
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
MeSH Terms: interventions — tislelizumab; Azacitidine; Lenalidomide; Etoposide; pegaspargase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TALE regimen (Experimental): tislelizumab plus azacytidine and lenalidomide
  Interventions: Drug: tislelizumab, azacytidine, lenalidomide
- TEPA regimen (Experimental): tislelizumab plus etoposide and pegaspargase
  Interventions: Drug: tislelizumab, etoposide, pegaspargase

INTERVENTIONS:
Drug: tislelizumab, azacytidine, lenalidomide — tislelizumab, 200mg, iv, day 1, every 21 days.
  azacytidine, 75mg/m2, ih, days 1-7, every 21 days.
  lenalidomide, 25mg, po, days 1-14, every 21 days.
  Other Names: Tileilizhu Dankang
  Arms: TALE regimen
Drug: tislelizumab, etoposide, pegaspargase — tislelizumab, 200mg, iv, day 1, every 21 days.
  etoposide, 100mg, iv, days 1-3, every 21 days.
  pegaspargase, 2000U/m2, day 1, every 21 days
  Other Names: Tileilizhu Dankang
  Arms: TEPA regimen

SUMMARY:
Natural killer/T-cell lymphoma (NKTCL) patients with relapsed/refractory disease had very poor outcome. Anti-PD-1 antibody showed promising results in response, but but the complete remission rate of was low. Some anti-PD-1 antibody based regimen showed higher and deeper response in NKTCL patients.

DETAILED DESCRIPTION:
About 20-30% of early-stage patients and 40-60% of late-stage NKTCL patients will experience disease relapse and refractory disease, and the median survival time of relapsed patients is about 6 months. PD-1 antibody is an effective drug for the treatment of patients with relapsed/refractory NKTCL, but the response rate and complete remission rate of monotherapy are low. How to improve the prognosis of patients is an important way to try combination therapy. In this study, we aim to explore the effectiveness and safety of a novel anti-PD-1 antibody, tislelizumab, in combination with different drugs (tislelizumab plus azacytidine and lenalidomide, or tislelizumab plus etoposide and pegaspargase) to treat refractory NK/T.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy histopathology, immunohistochemistry and EBER test meet ing the WHO 2016 diagnostic criteria for NK/T cell lymphoma.
2. With progressive disease after asparaginase-based combined chemotherapy
3. Have experienced multiple courses of PD-1/PD-L1 treatment with non-responsive or progressive disease.
4. PET/CT or CT/MRI with at least one measurable lesion or objectively evaluable lesion.
5. General ECOG score 0-3 points.
6. The laboratory examination within 1 week before enrollment meets the following conditions:

   Blood routine: Hb>80g/L, PLT>50×109/L. Liver function: ALT, AST, TBIL ≤ 2 times the upper limit of normal. Renal function: Cr is normal. Blood coagulation test: plasma fibrinogen ≥1.0g/L. Heart function: LVEF≥50%, ECG did not indicate any acute myocardial infarction, arrhythmia, or atrioventricular block of degree I or more.
7. Signed informed consent form.
8. Voluntarily comply with research protocols, follow-up plans, laboratory and auxiliary examinations.

Exclusion Criteria:

1. Patients with a history of pancreatitis (only patients who are planning to undergo PD1 combined with pegaspargase are excluded).
2. Severe infections require ICU treatment.
3. Combined HCV or HIV infection. Patients with HBV infection who receive antiviral treatment at the same time will not be excluded.
4. There are serious complications such as fulminant DIC.
5. Impairment of important organ functions: such as respiratory failure, chronic congestive heart failure with NYHA grade ≥2, decompensated liver or kidney insufficiency, hypertension and diabetes that cannot be controlled despite active treatment, nearly 6 years old There were cardio-cerebrovascular thrombotic or hemorrhagic events within months.
6. Pregnant and lactating women.
7. Have a history of autoimmune diseases, have disease activity in the past 6 months, and are still receiving oral immunosuppressive therapy within the past three months, and the daily dose of oral prednisone is greater than 10 mg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Week 12 +/-7 days
  The overall response rate will be assessed on Week 12

SECONDARY OUTCOMES:
Complete response rate | Week 12 +/-7 days
  The complete response rate will be assessed on Week 12
Progression free survival | 1-year
  Progression free survival is the time from entry onto the treatment until lymphoma progression or death of any reason.
Overall survival | 1-year
  Overall survival is defined as the time from entry onto the treatment until death of any reason
Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | Treatment-Related Adverse Events will be assessed and graded by NCI CTCAE v5.0.
  From day 1 of each course of chemotherapy to the 3 months after the last dose of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, MD, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No